CLINICAL TRIAL: NCT01237028
Title: Additive Renoprotective Effects of Oral Calcitriol in IgA Nephropathy Patients Taking Renin-Angiotensin System Blockers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2010-0439
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral calcitriol (Experimental): Calcio®
  Interventions: Drug: Calcitriol
- placebo (No Intervention)

INTERVENTIONS:
Drug: Calcitriol — Calcitriol(1,25-dihydroxycholecalciferol, vitamin D3 analog)0.25 μg per day
  Arms: oral calcitriol

SUMMARY:
This study will help to show the efficacy of vitamin D and address the optimal strategy to minimize renal injury in IgAN patients.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven Ig AN patients aged 20-70 years
* Patients with residual proteinuria > 500 mg/g creatinine despite renin-angiotensin system blockade and adequate blood pressure control for more than 3 months
* Patients who give informed consent, and 4) estimated GFR >= 30 ml/min/1.73 m2.

Exclusion Criteria:

* patients < 20 years or > 70 years
* hypersensitivity to vitamin D analogs
* patients who need urgent dialysis
* hypercalcemia within 3 months (uncorrected serum calcium level > 10.2 mg/dL)
* clinical features of rapidly progressive glomerulonephritis
* life expectancy less than 24 months
* uncontrolled hypertension
* decompensated liver or lung disease
* symptomatic heart failure (NYHA class II-IV or LVEF < 40%)
* estimated GFR < 30 ml/min/1.73 m2.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
changes in proteinuria | random urine protein/creatinine ratio every 2month and 24hour urine protein every 6month
  comparison of proteinuria amount checked by random urine protein/creatinine and 24hour urine protein

SECONDARY OUTCOMES:
changes in serum creatinine | serum creatinine every 2month
  comparison of renal function checked by serum creatinine and calculated renal function by MDRD equation
changes in systolic blood pressure and diastolic pressure | check blood pressure at very first visit and every 2-month
  check systolic and diastolic blood pressure
changes in urinary biomarkers (angiotensinogen, angiotensin II, TGF-beat, IL-6, MCP-1, TNF-alpha) | every 6month
  urine marker check every 6month
changes in serum 25(OH)2D3, 1,25(OH)2D3, parathyroid hormone | every 6month
  serum marker check every 6month
changes in serum inflammatory markers (hsCRP, IL-6) | every 6month
  serum marker check every 6month

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Hyun Yoo, MD, Ph.D, Principal Investigator — Severance Hospital
Locations (7):
- South Korea (7):
  - National Health Insurance Corporation Ilsan Hospital, Goyang
  - Kwandong University Myongji Hospital, Goyang
  - Wongkwang University Sanbon Medical Center, Gunpo
  - CHA University Bundang Medical Center, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Ewha Womans University Medical Center, Seoul